CLINICAL TRIAL: NCT03296501
Title: Safety and Efficacy of Intraspinal Transplantation of Autologous ADRC in ALS Patients
Brief Title: Intraspinal Transplantation of Autologous ADRC in ALS Patients
Acronym: ADIPOSTEM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mossakowski Medical Research Centre Polish Academy of Sciences (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Anna Sarnowska, M.D., Ph.D., Mossakowski Medical Research Centre Polish Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPO/014/33/09/2015
Record Dates: First submitted 2017-09-21; First posted 2017-09-28 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; ADRC; adipose derived regenerative cells; intraspinal transplantation; mesenchymal cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous ADRC injection (Experimental)
  Interventions: Biological: Cell-based therapy of autologous adipose derived regenerative cells transplanted intraspinally and intrathecally in ALS patients

INTERVENTIONS:
Biological: Cell-based therapy of autologous adipose derived regenerative cells transplanted intraspinally and intrathecally in ALS patients — 3 injections of ADRC: 1 intraspinal and 2 intrathecal

SUMMARY:
The goal of our nonrandomized, open label study is to investigate the safety and efficacy of autologous adipose derived mesenchymal regenerative cells (ADRC) transplantation into the individuals with diagnosed amyotrophic lateral sclerosis (ALS). All enrolled patients will have a documented at least 3-months clinical and electrophisiological observation of ALS disease course prior to study enrollment. Each patient will recive 3 injections of ADRC every 3 months: an intraspinal injection followed by 2 subsequent intrathecal infusions. Safety, adverse events and efficacy will be confirmed by clinical, elecrophisiological ( EMG, MUNIX), neuroimmaging and spirometry together with functional (ALSFRS-R) and objective motor assesment (MRC and dynamometer).

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is an incurable disease of unknown etiology that in a short time leads to significant impairment of motor functions and death. The frequency of ALS is 4-8/100 000. Mostly it affects people between 40 and 70 years old, but it can occur at a younger age. Since the symptom onset is most frequently in the fifth or sixth decade, ALS is a huge economic burden for the society. There are many studies conducted to treat the disease and prevent it, but currently the medicine offers only one drug that can slow the appearance of disease symptoms but could not stop the progression. Yet, improvements in medical management, including nutrition and breathing, regularly increase patient survival - 50% of affected patients live at least 3 or more years after diagnosis; 20% live 5 years or more; and up to 10% will survive more than 10 years. The stem-cell-based therapies could be therefore a new waited strategy for ALS clinical treatment.

Since the clinical course of ALS may vary substantially between patients, we are planning to qualify them with a primarily established clinical course based on a detailed anamnesis and clinical assessment. The goal of our nonrandomized, open label study is to investigate the safety and efficacy of autologous adipose derived mesenchymal regenerative cells (ADRC) transplantation into the individuals with diagnosed amyotrophic lateral sclerosis. In order to select a group of 30 ALS patients for the ADRC treatment, approximately 50 ALS patients will be examined. All patients enrolled will have a documented at least 3-months clinical and electrophisiological observation of ALS disease course prior to study enrollment. Each patient will recive 3 injections of ADRC every 3 months: an intraspinal injection followed by 2 subsequent intrathecal infusions. Safety, adverse events and efficacy will be confirmed by clinical, elecrophisiological ( EMG, MUNIX), neuroimmaging and spirometry together with functional (ALSFRS-R) and objective motor assesment (MRC and dynamometer).

ELIGIBILITY:
Inclusion Criteria:

* clinically definite or probable ALS according to El Escorial criteria
* life expectancy of more than 1 year
* INR ≤2 before liposuction
* lack of treatment with immune-suppressants and/or corticosteroids within min. 20 days prior to recruitment
* constant riluzole treatment (50 mg/bid) throughout the study period
* compliance with treatment regimen e.g. will and possibility to attend check-up visits
* Polish citizens

Exclusion Criteria:

* primary haematological disease, including hypercoagulable states
* Presence of comorbidity that would stand in the way of neurosurgical treatment-
* previous history of a spinal-cord surgery at the clinically affected level
* previous/current history of neoplasm or comorbidity that could impact upon patient's survival
* PEG
* pregnancy /lactation
* noninvasive/invasive mechanical ventilation at time of recruitment
* alcohol abuse, cocaine amphetamine, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10-13 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Functional progression rate | 3 months
  Delta ALS Functional Rating Scale (ALSFRS-R)/month

SECONDARY OUTCOMES:
Electrophisiological progression rate | 3 months
  electromyography (EMG)/ Motor unit number index (MUNIX)

OTHER OUTCOMES:
Respiratory insufficiency estimation | 3 months
  Forced Vital Capacity (FVC)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuzma-Kozakiewicz M, Marchel A, Kaminska A, Gawel M, Sznajder J, Figiel-Dabrowska A, Nowak A, Maj E, Krzesniak NE, Noszczyk BH, Domanska-Janik K, Sarnowska A. Intraspinal Transplantation of the Adipose Tissue-Derived Regenerative Cells in Amyotrophic Lateral Sclerosis in Accordance with the Current Experts' Recommendations: Choosing Optimal Monitoring Tools. Stem Cells Int. 2018 Aug 12;2018:4392017. doi: 10.1155/2018/4392017. eCollection 2018. PMID 30158984